CLINICAL TRIAL: NCT03106194
Title: Case Management in Hepatitis C Virus Infected People Who Inject Drugs in Belgium
Brief Title: Case Management in HCV Infected PWID
Acronym: CM-HCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other); CAD Limburg (Unknown)
Responsible Party: Principal Investigator, Geert Robaeys, prof. dr., Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ZOL-CM-HCV
Record Dates: First submitted 2017-02-22; First posted 2017-04-10 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Drug Abuse, Intravenous
MeSH Terms: conditions — Substance Abuse, Intravenous | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- history of injection drug use (Other): Men and women ≥ 18 years old with a history of injection drug use, enrolled in the opiate substitution program of CAD Limburg.
  Case management
  Interventions: Other: case management

INTERVENTIONS:
Other: case management

SUMMARY:
To study the impact of case management on the outcome of the care of chronic hepatitis C in people who inject drugs (PWID). By creating the function of case manager, the investigators will target all the barriers to care of the HCV care continuum. Partial objectives are to measure the impact of case management on the uptake for screening, the uptake and outcome of treatment, and the rate of reinfection.

DETAILED DESCRIPTION:
Hepatitis C virus infection (HCV) is nowadays one of the leading causes of chronic liver disease, with prevalence of liver cirrhosis still increasing. The hepatitis C virus (HCV) is primarily transmitted through blood-to-blood contact. In the Western world, overall prevalence of HCV antibodies is low. In Belgium, prevalence of HCV in the general population is estimated around 1% by expert opinion. However, in high-risk populations prevalence of HCV increases. Data for HCV antibody prevalence in Belgium show rates of 60-80% in people who inject drugs (PWID). Populations at increased risk of HCV infection include:

* PWID
* recipients of infected blood products or invasive procedures in health-care facilities with inadequate infection control practices (western world: before 1992)
* children born to mothers infected with HCV
* people with sexual partners who are HCV-infected
* people with HIV infection
* prisoners or previously incarcerated persons
* people who have used intranasal drugs
* people who have had tattoos or piercings

Based on international guidelines, the Belgian Association for the Study of the Liver (BASL) recommends targeted screening for these populations to assess HCV prevalence. This is not yet executed in Belgium, despite the severe health and economic burden accompanied with chronic hepatitis C virus infection (CHC). In response to this lacuna in the Belgium health care, the "Hepatitis C Plan (2014-2019)" was developed. This action plan aims to improve the following goals:

* Uptake for screening in high-risk populations
* Creation of a national systematic screening procedure
* Development of an HCV expertise network to improve care and linkage-to-care Furthermore, in April of 2015 the federal government of Belgium distributed a pact with the pharmaceutical industry, called "The Future Pact". This pact between industry and government focuses on accessibility to care, specifically for high-risk groups. Goals are to create a national registry for therapy and develop patient support programs, next to the expansion of reimbursement of therapy for HCV infection in fibrosis stadium II. However, despite the international guidelines and despite the strategic aims in the Hepatitis C plan and the Future Pact, no specific actions are described, and screening is not systematically executed in high-risk groups in Belgium.

The importance of this screening cannot be underestimated as HCV is now curable, with success rates of 60-100% according to other associated factors (e.g. use of direct acting antivirals (DAAs), severity of liver disease, HCV genotype, resistance). Furthermore, different studies state that treatment of patients with CHC in an early stage has the potential to be cost-effective, as hospitalization costs after development of liver disease far exceed the cost of antiviral therapy. Nonetheless, treatment uptake also remains low.

One of the reasons why PWIDs were excluded from treatment in the past was stigmatization based on greater risk of reinfection. Latest studies show low rates of reinfection among PWID, even with continued injection drug use during and after treatment. The pooled HCV reinfection risk was 2.4 per 100 person years, combined for six studies, across the UK, Australia, the Netherlands and Greece, suggesting that HCV treatment should not be withheld due to concerns about reinfection alone. However, with ongoing risk behaviour, current guidelines recommend monitoring with annual HCV RNA assessments. Furthermore, data from the National Scottish Hepatitis C Clinical Database show that an increasing significant minority of PWID continue to inject post-SVR at an intensity which leads to either hospitalisation or death and increased risk of reinfection. Thus, harm reduction and counselling remain necessary.

With this trial, the investigators want to evaluate a possible approach to reach the different goals defined in the Hepatitis C plan and the future pact. The investigators will study the impact of case management on the outcome of care for HCV infected PWID in Belgium.

ELIGIBILITY:
Inclusion criteria

* ≥ 18 years of age
* History of injection drug use with substitution program
* Written informed consent obtained

Exclusion criteria

* Possible acute HCV infection within the previous 6 months defined by one of the following: acute hepatitis symptoms, ALT ≥ 10x ULN, negative or unknown HCV antibody status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Uptake for screening (%) | screening
  percentage of clients screened in relation to number of clients in follow-up at CAD
Uptake for treatment assessment (%) | day 1
  percentage of HCV positive clients who attented a hepatology consultation in relation of total of HCV positive clients
Uptake for treatment (%) | day 1
  percentage of HCV positive clients who started treatment in relation of total of HCV positive clients needing treatment
Compliance to therapy (%) | up to three years
  percentage of patients reaching end-of treatment response, who present at the consultation, in relation to total patients in treatment
Rate of sustained viral response (SVR) (%) | up to three years
  percentage of patients who clear the hepatitis C virus in relation to total patients treated
Rate of reinfection (%) | up to three years
  percentage of patients who get reinfected with HCV in relation to total cured patients

CONTACTS AND LOCATIONS:
Overall Officials: Geert Robaeys, prof. dr., Principal Investigator — Hasselt University; Rob Bielen, drs., Study Chair — Hasselt University
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Busschots D, Bielen R, Koc OM, Heyens L, Dercon E, Verrando R, Janssens F, Van den Bergh L, Van Lint P, Bruckers L, Nevens F, Robaeys G. On-site testing and case management to improve hepatitis C care in drug users: a prospective, longitudinal, multicenter study in the DAA era. BMC Public Health. 2021 Aug 20;21(1):1574. doi: 10.1186/s12889-021-11608-9. PMID 34416867